CLINICAL TRIAL: NCT04775745
Title: A Phase I, Multicenter, Open-Label, Dose-escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Clinical Activity of Orally Administered LP-168 in Subjects With Relapsed or Refractory B-cell Malignancies.
Brief Title: Study of Oral Administration of LP-168 in Patients With Relapsed or Refractory B-cell Malignancies.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newave Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LP-168-US-I01
Record Dates: First submitted 2021-02-22; First posted 2021-03-01 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: CLL/SLL; Waldenstrom Macroglobulinemia; Follicular Lymphoma; Diffuse Large B Cell Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Hairy Cell Leukemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Hairy Cell

STUDY DESIGN:
Intervention Model Description: A classic "3+3" design will be used to establish the dose-limiting toxicity (DLT), MTD, and RP2D. Three to six subjects per treatment cohort will be assigned to receive sequentially higher oral doses of LP-168 on a once or twice daily schedule for 28 days (a "Cycle"), starting at a dose of 100 mg/day. Once all subjects in a given cohort have reached Cycle 1 Day 28, these data will be reviewed by the Safety Review Committee (SRC) for decisions on dose escalation for a new dose cohort. Subjects will receive once-daily or twice-daily oral dose of LP-168 until disease progression, unacceptable toxicity, or a clinical observation satisfying another criterion for withdrawal from treatment is noted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Phase (Experimental): Three to six subjects per treatment cohort will be assigned to receive sequentially higher oral doses of LP-168 on a once or twice daily schedule for 28 days, starting at a dose of 100 mg/day.
  Interventions: Drug: LP-168
- Dose Expansion Phase (Experimental): Additional subjects will be recruited to further explore the safety, tolerability, PK, and efficacy in specific subject subgroups.
  Interventions: Drug: LP-168

INTERVENTIONS:
Drug: LP-168 — For the dose escalation phase, LP-168 will be given once or twice daily at the following dose levels:100 mg QD,150 mg QD, 100 mg BID, 300 mg QD, 150 mg BID, 450 mg QD, 225 mg BID, 600 mg QD, 800 mg QD, and 1000 mg QD.
  Arms: Dose Escalation Phase
Drug: LP-168 — For the dose expansion phase, subjects will receive once or twice daily dose of LP-168 at the Recommended Phase 2 Dose (RP2D). The RP2D may be as high as the MTD and will be determined following evaluation of Phase I Dose Escalation results.
  Arms: Dose Expansion Phase

SUMMARY:
This is a phase I, multi-center, open-label, dose-escalation study to evaluate the safety, tolerability, pharmacokinetics and clinical activity of LP-168 in subjects with relapsed or refractory B-cell malignancies. LP-168 is a small molecule inhibitor.

DETAILED DESCRIPTION:
The primary objectives for the study are to assess the safety and tolerability profile, determine the maximum tolerated dose (MTD), and/or the recommended Phase 2 dose (RP2D) of LP-168 administered once or twice daily as a single agent dosed orally in adult subjects with relapsed/refractory B-cell Malignancies (CLL/SLL, WM, FL, MCL, MZL, DLBCL, HCL); and to characterize the pharmacokinetics (PK) profile of LP-168 in adult subjects with relapsed/refractory B-cell Malignancies (CLL/SLL, WM, FL, MCL, MZL, DLBCL, HCL).

Secondary objectives of the study are to evaluate preliminary efficacy regarding the effect of LP-168 on progression-free survival (PFS), objective response rate (ORR), and duration of response (DOR) in adult subjects with relapsed/refractory B-cell Malignancies (CLL/SLL, WM, FL, MCL, MZL, DLBCL, HCL).

Once the MTD is declared and the RP2D is established, additional subjects will be enrolled in a cohort expansion phase (Phase 1b).

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for study participation if he/she meets the following criteria:

* Subjects are eligible with B-cell malignancies, WM, FL, MCL, MZL, DLBCL, HCL, CLL, SLL, based upon 2016 updated WHO classification. Those subjects with WM, FL, MCL, DLBCL, or HCL must have received at least 2 prior systemic therapies.
* Low-grade B-cell lymphomas as follicular Grade 1, 2, or 3A, marginal zone or small lymphocytic lymphoma.
* Subject must have adequate coagulation, renal, and hepatic function, per local laboratory reference ranges at Screening as follows:

  * Activated partial thromboplastin time (APTT) and prothrombin time (PT) not to exceed 1.5 × ULN
  * Calculated creatinine clearance (CrCl) ≥ 60 mL/min using 24-hour CrCl OR Cockcroft-Gault formula.
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 1.5 ×ULN; Bilirubin ≤ 1.5 × ULN (except subjects with Gilbert's Syndrome, who may have a bilirubin > 1.5 × ULN, per discussion between the Investigator and the Medical Monitor).
* Subjects must have adequate bone marrow independent of growth factor support per local laboratory reference range at screening as follows:

  * Absolute Neutrophil Count (ANC) ≥1000/uL;
  * An exception is for subjects with an ANC<1000/uL and bone marrow heavily infiltrated with underlying disease (approximately 60% or more) may use growth factor to achieve the ANC eligibility criteria per discussion between the Investigator and the Medical Monitor.
  * Platelet count ≥ 50,000/µL - OR - Platelet count ≥ 20,000/ µL if thrombocytopenia is clearly due to CLL disease under study (per Investigator discretion)
  * Hemoglobin ≥8.0g/dL, and can be achieved by transfusion

Exclusion Criteria:

A subject will not be eligible for study participation if he/she meets any of the following criteria.

* Subject has received any of the following therapies within 14 days or 5 half-lives (whichever is shorter) prior to the first dose of study drug, or has not recovered to ≤ Grade 1 clinically significant adverse effect(s)/toxicity(s) of the previous therapy (other than alopecia):

  * Any anti-cancer therapy including chemotherapy, biologic or immunotherapy, radiotherapy, etc;
  * Any investigational therapy, including targeted small molecule agents.
  * For CLL subjects who come off BCR antagonists (BTK inhibitors, PI3K inhibitors, etc.) treatment, allow washout for 2 days as these subjects progress quickly after treatment discontinuation and then remain eligible (steroids may be given during these two days to allow disease control).
* Subjects who require immediate cytoreduction. However, subjects may receive up to two days of steroids for symptoms of impending organ impairment and remain eligible.
* Subject has received the following medications or therapies within 7 days prior to the first dose of study drug:

  * Steroid therapy (at dosages equivalent to prednisone >20 mg/day) for anti-neoplastic intent (except as noted in exclusion criteria #3);
  * Cytochrome P450, family 3, subfamily A (CYP3A4) strong inhibitors and strong CYP2C8 inducers/inhibitors.
  * Potent CYP3A4 inducers such as rifampin, carbamazepine, phenytoin, and St. John's wort.
* Subjects require treatment with systemic acid-reducing agents including H-2-receptor antagonists and proton pump inhibitors with the following exceptions:

  * Proton pump inhibitors should be discontinued at least 7 days prior and held throughout the study
  * If concurrent use of an H2 blocking agent is necessary, it must be administered only between 2 and 3 hours after the dose of LP-168. If not taken during this time, the dose of H2 blocking agents should not be taken again until 2-3 hours after the next dose of LP-168.
  * If concurrent use of a local antacid is necessary, it must be administered 2 or more hours before and/or 2 or more hours after the dose of LP-168.
* Subject has significant screening electrocardiogram (ECG) abnormalities including. 2nd degree AV block type II 3rd degree block, Grade 2 or higher bradycardia, and corrected QT interval (QTc) ≥ 480ms.
* Serum amylase > 1.5 × ULN or serum lipase > 1.5 × ULN.
* Subject has any history of Richter's transformation for Phase 1a portion of the trial.
* Subjects who have undergone autologous/allogeneic hematopoietic stem cell transplantation (HSCT) therapy within 90 days of the first dose of LP-168, or patients on immunosuppressive therapy post-HSCT at the time of Screening, or currently with clinically significant graft-versus-host disease (GVHD) as per treating physician (Patients in relapse after allogeneic transplantation must be off treatment with systemic immunosuppressive agents for at least 4 weeks. The use of topical steroids and/or up to 20 mg/day prednisone or equivalent systemic steroids for ongoing GVHD is permitted.
* Subject has a history of other active malignancies other than B-cell malignancies within the past 3 years prior to study entry, with the exception of:

  * Adequately treated in situ carcinoma of the cervix uteri;
  * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
  * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.
* Subject requires anticoagulation with Warfarin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to 24 months, each cycle is 28 days
  When more than 1 DLT occurs in ≤ 6 subjects in a dosing cohort, dose escalation will be stopped and this dose level will be identified as the non-tolerated dose. Doses between the non-tolerated dose and the preceding lower dose, where ≤ 1 DLT occurred, may be explored to more precisely define the MTD.
Recommended Phase 2 dose (RP2D) | Up to 24 months, each cycle is 28 days
  The RP2D may be as high as the MTD or a lower dose and will be selected in discussion with the Investigators and the Sponsor based on longer term safety data, preliminary efficacy data, and PK data.
Pharmacokinetic (PK) profile of LP-168 | At Cycle 1: Day 1, Day 2, Day 8, Day 9, Day 15, Day 22, Day 28; At Cycle 3: Day 28; At Cycle 6 Day 28; (each cycle is 28 days)
  Maximum Plasma Concentration [Cmax]
Pharmacokinetic (PK) profile of LP-168 | At Cycle 1: Day 1, Day 2, Day 8, Day 9, Day 15, Day 22, Day 28; At Cycle 3: Day 28; At Cycle 6 Day 28; (each cycle is 28 days
  Area Under the Curve [AUC]
Pharmacokinetic (PK) profile of LP-168 | At Cycle 1: Day 1, Day 2, Day 8, Day 9, Day 15, Day 22, Day 28; At Cycle 3: Day 28; At Cycle 6 Day 28; (each cycle is 28 days
  Time at Maximum Concentration [Tmax]

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 24 months, each cycle is 28 days
  PFS is measured from the time of first study drug administration until the first date that recurrent or progressive disease is objectively documented.
Objective Response Rate (ORR) | Up to 24 months, each cycle is 28 days
  ORR is defined as the sum of complete response (CR) and partial remission rates.
Duration of Response (DOR) | Up to 24 months, each cycle is 28 days
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (which is first recorded) until the first date that recurrent or progressive disease is objectively documented

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Duke Univerisity, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No